CLINICAL TRIAL: NCT06859541
Title: Culturally Adapted Play-Based Behavioural Intervention Among Children With Autism Spectrum Disorder in Semi-Rural Tamil Nadu: A Randomized Controlled Trial
Brief Title: Culturally Adapted Play-Based Behavioural Intervention for Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saveetha University (Other)
Responsible Party: Principal Investigator, Madhanraj Sekar, Principal Investigator, Saveetha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 322/07/2024/ISRB/UGSR/SCPT
Record Dates: First submitted 2025-02-23; First posted 2025-03-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Adaptive Behaviour; Autism Spectrum Disorder; Behaviour Therapy; Play Therapy; Semi-Rural Tamil Nadu
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally Adapted Play-Based Behavioural Intervention Group (Experimental): The Culturally Adapted Play-Based Behavioural Intervention (PPBI) incorporated traditional Tamil games and folk storytelling to enhance social awareness, emotional regulation, and language development. Over 12 weeks, the program progressed through key developmental areas:
  Weeks 1-2: Focused on engagement and communication through interactive activities.
  Weeks 3-4: Developed sensory and motor skills using creative play. Weeks 5-6: Strengthened language and expression with role-playing and storytelling.
  Weeks 7-8: Addressed emotional regulation through structured games and music therapy.
  Weeks 9-10: Encouraged social interaction with group play and problem-solving tasks.
  Weeks 11-12: Emphasized real-world application through community-based activities.
  Interventions: Behavioral: Culturally Adapted Play-Based Behavioural Intervention
- Applied Behaviour Analysis (Active Comparator): The Applied Behaviour Analysis (ABA) program was structured into progressive stages, each targeting specific behavioral improvements.
  Weeks 1 & 2: Introduced structured learning techniques, focusing on basic commands, eye contact training, and reinforcement strategies, such as reward-based motivation systems.
  Weeks 3 & 4: Emphasized early communication development, incorporating imitation exercises, visual schedules, and simple verbal response training.
  Weeks 5 & 6: Implemented behavior modification techniques, including token-based reinforcement, redirection methods, and gradual shaping of desired behaviors.
  Weeks 9 & 10: Focused on independent task execution, covering self-care routines such as dressing, eating, and personal hygiene, with structured multi-step guidance.
  Weeks 11 & 12: Aimed at generalizing learned behaviors, ensuring that children could apply their skills effectively in home, school, and social environments.
  Interventions: Behavioral: Applied Behaviour Analysis

INTERVENTIONS:
Behavioral: Culturally Adapted Play-Based Behavioural Intervention — The Culturally Adapted Play-Based Behavioural Intervention (PPBI) integrates traditional Tamil games and folk storytelling to enhance social, emotional, and communication skills in children with Autism Spectrum Disorder (ASD). This 12-week structured program focuses on engagement, motor development, language, emotional regulation, social interaction, and real-world skill application, making it a culturally relevant and accessible intervention for improving adaptive behaviours.
  Arms: Culturally Adapted Play-Based Behavioural Intervention Group
Behavioral: Applied Behaviour Analysis — The ABA-based program utilized structured techniques focused on positive reinforcement, imitation training, guided communication, and step-by-step skill-building. The primary goal was to reduce problem behaviors while reinforcing desirable social and communication skills. Parents and teachers were provided with structured training on how to apply ABA strategies consistently at home and school.
  Arms: Applied Behaviour Analysis

SUMMARY:
This study compared Culturally Adapted Play-Based Behavioural Intervention (PPBI) and Applied Behaviour Analysis (ABA) for children with Autism Spectrum Disorder (ASD) in semi-rural Tamil Nadu through a double-blinded randomized controlled trial with 56 participants.

The PPBI approach integrated traditional Tamil games such as Paandi (hopscotch), Kuzhi Thanda (hole-and-peg game), and Paramapadham (snakes and ladders) to encourage social interaction, cooperative play, motor skill development, and emotional self-regulation. Activities were structured to progress through various developmental goals, including turn-taking, gesture-based communication, sensory-motor coordination, language expression, peer collaboration, and real-life scenario practice. Additionally, storytelling, music-based play, and movement exercises were included to enhance communication and social awareness.

On the other hand, the ABA-based program utilized structured techniques focused on positive reinforcement, imitation training, guided communication, and step-by-step skill-building. The primary goal was to reduce problem behaviors while reinforcing desirable social and communication skills. Parents and teachers were provided with structured training on how to apply ABA strategies consistently at home and school.

DETAILED DESCRIPTION:
This research investigated the effectiveness of a Culturally Adapted Play-Based Behavioural Intervention (PPBI) in comparison to Applied Behaviour Analysis (ABA) for improving behavioral and social skills in children diagnosed with Autism Spectrum Disorder (ASD) in a semi-rural region of Tamil Nadu. Recognizing the challenges children with ASD face in communication, emotional regulation, and social interaction, the study aimed to explore whether an intervention rooted in traditional play-based methods could provide better engagement and outcomes.

A double-blinded randomized controlled trial was conducted, involving 56 children between the ages of 8 and 12, who were evenly divided into two groups: PPBI and ABA. Both programs ran five days a week over a 12-week period, with behavioral assessments conducted using the Strengths and Difficulties Questionnaire (SDQ). Parents and teachers provided input at multiple time points to capture changes in home and school environments. The research took place at Aadhuraa Special School in Kanchipuram, Tamil Nadu, ensuring the intervention was delivered in a setting that aligned with the children's cultural background.

Intervention Details:

The PPBI approach integrated traditional Tamil games such as Paandi (hopscotch), Kuzhi Thanda (hole-and-peg game), and Paramapadham (snakes and ladders) to encourage social interaction, cooperative play, motor skill development, and emotional self-regulation. Activities were structured to progress through various developmental goals, including turn-taking, gesture-based communication, sensory-motor coordination, language expression, peer collaboration, and real-life scenario practice. Additionally, storytelling, music-based play, and movement exercises were included to enhance communication and social awareness.

On the other hand, the ABA-based program utilized structured techniques focused on positive reinforcement, imitation training, guided communication, and step-by-step skill-building. The primary goal was to reduce problem behaviors while reinforcing desirable social and communication skills. Parents and teachers were provided with structured training on how to apply ABA strategies consistently at home and school.

ELIGIBILITY:
Inclusion Criteria:

Children aged 8 to 12 years diagnosed with Autism Spectrum Disorder (ASD) (mild to moderate severity).

Diagnosis confirmed using the Indian Scale for Assessment of Autism (ISAA). Classified as Level I to III in the Communication Function Classification System.

Attended regular sessions throughout the 12-week intervention. Parents or guardians provided informed consent and participated in training sessions.

Completion of behavioral assessments using the Strengths and Difficulties Questionnaire (SDQ).

Exclusion Criteria:

Children with severe ASD or comorbid neurological/psychiatric disorders. Those undergoing intensive behavioral therapy or other structured interventions.

Children with uncorrected sensory impairments (e.g., hearing or visual deficits) that could interfere with intervention activities.

Families unable to commit to the full 12-week study period.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | Baseline, 4th week, 8th week, 12th week
  The 25 item Strengths and Difficulties Questionnaire (SDQ) measures behavioral and emotional function. These 25 items are divided into 5 subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. The Strengths and Difficulties Questionnaire is scored on a 3-point Likert-type scale, with total scores (excluding the prosocial scale) ranging from 0 to 40. Higher scores reflect greater behavioral and emotional difficulties and lower scores reflects lesser behavioural and emotional difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Madhanraj S, Principal Investigator — Tutor; Jeevarathinam Thirumalai, Principal Investigator — Saveetha College of Physiotherapy, Saveetha Institute of Medical and Technical Sciences
Locations (1):
- Aadhuraa Special School, Kanchipuram, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kumar A, Bhattacharya S. Unveiling autism spectrum disorder in South East Asia through a public health Lens. Front Child Adolesc Psychiatry. 2024 Dec 4;3:1489269. doi: 10.3389/frcha.2024.1489269. eCollection 2024. PMID 39816604
- [Result] Chauhan A, Singh M, Jaiswal N, Agarwal A, Sahu JK, Singh M. Prevalence of Cerebral Palsy in Indian Children: A Systematic Review and Meta-Analysis. Indian J Pediatr. 2019 Dec;86(12):1124-1130. doi: 10.1007/s12098-019-03024-0. Epub 2019 Jul 13. PMID 31300955
- [Result] Dey I, Chakrabarty S, Nandi R, Shekhar R, Singhi S, Nayar S, Ram JR, Mukerji S, Chakrabarti B. Autism community priorities in diverse low-resource settings: A country-wide scoping exercise in India. Autism. 2024 Jan;28(1):187-198. doi: 10.1177/13623613231154067. Epub 2023 Mar 31. PMID 36999343
- [Result] Leaf JB, Leaf R, McEachin J, Taubman M, Ala'i-Rosales S, Ross RK, Smith T, Weiss MJ. Applied Behavior Analysis is a Science and, Therefore, Progressive. J Autism Dev Disord. 2016 Feb;46(2):720-31. doi: 10.1007/s10803-015-2591-6. PMID 26373767
- [Result] Deniz E, Francis G, Torgerson C, Toseeb U. Parent-mediated play-based interventions to improve social communication and language skills of preschool autistic children: A systematic review and meta-analysis protocol. PLoS One. 2022 Aug 15;17(8):e0270153. doi: 10.1371/journal.pone.0270153. eCollection 2022. PMID 35969530